CLINICAL TRIAL: NCT06680245
Title: Effect of Mitomycin-C on the Outcomes of Patients Receiving Ahmed Glaucoma Valve Implantation Surgery
Acronym: MMC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Enitan Sogbesan, Doctor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16370
Record Dates: First submitted 2024-05-27; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma
Keywords: Refractory Glaucoma; Intraocular Pressure; Ahmed Glaucoma Valve; Mitomycin-C; Glaucoma Surgery
MeSH Terms: conditions — Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: The study design is a parallel-armed clinical superiority randomized trial. The study participants will be blinded to the use of the mitomycin-c with the Ahmed valve implant. Participants will be randomly allocated to either the experimental group using mitomycin-c injections or the control group receiving no intervention. The trial will be conducted at the Hamilton Regional Eye Clinic at St. Joseph's Healthcare Hamilton to maintain standardization of care and follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: There will be no blinding of the ophthalmologist to participant's study group as they will need the information to execute the correct intervention. The type of treatment received (mitomycin-C or no intervention) will be blinded for the patient, and all patients will be asked at the last follow-up visit which treatment location they felt they received. This data will be used to assess the level of treatment masking. The success of blinding will be calculated using Bang's Blinding Index. The person performing statistical analysis will be blinded to the intervention groups. The groups will be coded and the analyst will be unaware of which group receives mitomycin-C or no intervention with the Ahmed valve implant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mitomycin-C Treatment (Experimental): The intervention aims to assess the efficacy of Mitomycin-C in preventing postoperative hypertensive phases by inhibiting fibroblast proliferation around the surgical site. Patients in this arm will receive a 0.2 mg/mL Mitomycin-C injection into the sclera during Ahmed Glaucoma Valve implantation surgery. The total volume of the injection will be 1 mL, administered once intraoperatively.
  Interventions: Drug: Mitomycin c
- Control (No Intervention): Patients in this arm will undergo the Ahmed Glaucoma Valve implantation surgery without the addition of Mitomycin-C. This group serves as a control to evaluate the effects of the Ahmed Valve alone in managing intraocular pressure in patients with refractory glaucoma. Postoperative care remains consistent with the experimental group, involving the same regimen of topical antibiotics and steroids.

INTERVENTIONS:
Drug: Mitomycin c — Patients needing Ahmed valve implants to control intraocular pressures will be eligible. Eligible patients who consent will be randomized to receive either mitomycin-C or no intervention during implant surgery. Screening visits occur one week before surgery to assess eligibility and take baseline measurements (visual acuity, IOP, anterior chamber reaction). On surgery day, patients register at SJHH King Campus and undergo randomization. IOP is measured using a tonopen in the OR. An experienced glaucoma specialist performs the surgery, injecting 0.2 mg/ml mitomycin-C into the sclera for the experimental group, while the control group receives no intervention. The area is irrigated with 40mL balanced salt solution before implant insertion. Post-operative care includes topical antibiotics and steroids for six weeks, with follow-ups at 1 and 2 weeks, and 1, 3, 6, and 12 months to monitor visual acuity, IOP, anterior chamber reaction, complications, and additional glaucoma medications.
  Arms: Mitomycin-C Treatment

SUMMARY:
The goal of this clinical trial is to determine if the intraoperative application of Mitomycin-C can enhance the outcomes of Ahmed Glaucoma Valve (AGV) implantation in treating refractory glaucoma. This study is conducted among adult patients diagnosed with refractory glaucoma, a condition characterized by uncontrolled intraocular pressure despite the use of maximum tolerated medical therapy and previous surgical interventions. The main questions it aims to answer are:

Does intraoperative Mitomycin-C reduce postoperative intraocular pressure more effectively than surgery without it? Does Mitomycin-C reduce the occurrence of postoperative complications such as hypertensive phases?

Researchers will compare the experimental group receiving Mitomycin-C during AGV implantation to the control group undergoing AGV implantation without Mitomycin-C to see if the treatment leads to lower intraocular pressure and fewer surgical complications.

Participants will:

* Undergo baseline assessment including eye examination and measurement of intraocular pressure.
* Be randomly assigned to receive either the Mitomycin-C treatment or no intervention during their scheduled AGV implantation surgery.
* Attend follow-up visits at 1 week, 1 month, 3 months, 6 months, and 12 months post-surgery to assess intraocular pressure, visual acuity, and any postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (OAG); including ocular hypertension, pigmentary dispersion syndrome and pseudoexfoliation syndrome
* Participant must be over 18 years of age
* IOP > 16mmHg on at least two consecutive occasions separated by one month
* Two sighted eyes with visual acuity of 20/200 or better
* Informed consent from patient

Exclusion Criteria:

* Diagnosis of secondary OAG (aside from pigmentary and pseudoexfoliation glaucoma) or narrow angle glaucoma
* Previous incisional glaucoma surgery
* Incisional glaucoma surgery scheduled within 1 year of intervention
* Corneal disease affecting visualization of anterior chamber of the eye
* Treatment or plan to treat with topical or systemic steroids
* Previous laser treatments (selective laser trabeculoplasty or Argon laser trabeculoplasty)
* Other eye disorders or surgical procedures (ie retinal detachment) that may influence the results of glaucoma surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Intraocular Pressure assessed using the Goldmann applanation tonometer | Baseline to 1-year follow-up visit
  The percentage decrease in intraocular pressure (IOP) from baseline will be calculated and compared between the two groups from baseline to 1-year follow-up. It will be measured using the Goldmann applanation tonometer and performed at approximately the same time of the day to account for diurnal variation. Two measurements will be averaged if the difference is less or equal to 2mmHg. If the difference is greater than 2mmHg, then three measurements will be taken and the median will be recorded. The baseline IOP will be the average of three different IOP values taken at different times of the day on at least two separate days within a period of a month. In this study, the baseline IOP will be the average IOP of previous IOP measurement and the day of surgery.

SECONDARY OUTCOMES:
Number of Glaucoma Medications assessed by reviewing of patient medication records | Baseline to 1-year follow-up visit
  Changes in the number of glaucoma medications need per patient in each group will be compared using observations and by reviewing patient medication records from baseline to 1-year follow-up. This outcome will assess whether the intervention affects the number of prescribed glaucoma medications for the patients.
Visual Acuity assessed using the Snellen chart. | Baseline to 1-year follow-up visit
  Changes in visual acuity from baseline to 1-year follow-up will be measured using the Snellen chart. This outcome will assess whether the intervention affects the overall visual function of the patients.
Anterior Chamber Inflammation assessed using the Slit-lamp examination | Baseline to 1-year follow-up visit
  The anterior chamber inflammation at every post-operative visit will be compared to assess any complications during the surgery. This will be measured using the slit-lamp examination.
Progression to Surgical Therapy measured using clinical evaluation and surgical records. | Baseline to 1-year follow-up visit
  The progression to surgical therapy in each group will be compared from baseline to 1-year follow-up.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinreb RN, Aung T, Medeiros FA. The pathophysiology and treatment of glaucoma: a review. JAMA. 2014 May 14;311(18):1901-11. doi: 10.1001/jama.2014.3192. PMID 24825645
- [Background] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Background] Margolis KL, Rich EC. Open-angle glaucoma. Prim Care. 1989 Mar;16(1):197-209. PMID 2649902
- [Background] Sharts-Hopko NC, Glynn-Milley C. Primary open-angle glaucoma. Am J Nurs. 2009 Feb;109(2):40-7; quiz 48. doi: 10.1097/01.NAJ.0000345434.37734.ee. PMID 19299999
- [Background] Alasbali T, Alghamdi AA, Khandekar R. Outcomes of Ahmed valve surgery for refractory glaucoma in Dhahran, Saudi Arabia. Int J Ophthalmol. 2015 Jun 18;8(3):560-4. doi: 10.3980/j.issn.2222-3959.2015.03.22. eCollection 2015. PMID 26086008
- [Background] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Background] Riva I, Roberti G, Oddone F, Konstas AG, Quaranta L. Ahmed glaucoma valve implant: surgical technique and complications. Clin Ophthalmol. 2017 Feb 17;11:357-367. doi: 10.2147/OPTH.S104220. eCollection 2017. PMID 28255226
- [Background] Kurnaz E, Kubaloglu A, Yilmaz Y, Koytak A, Ozertrk Y. The effect of adjunctive mitomycin C in Ahmed glaucoma valve implantation. Eur J Ophthalmol. 2005 Jan - Feb 2005;15(1):27-31. doi: 10.5301/EJO.2008.210. PMID 28221428
- [Background] Luzu J, Baudouin C, Hamard P. The role of Ahmed glaucoma valve in the management of refractory glaucoma: Long-term outcomes and complications. Eur J Ophthalmol. 2021 Sep;31(5):2383-2389. doi: 10.1177/1120672120968733. Epub 2020 Nov 25. PMID 33238768
- [Background] Amoozgar B, Lin SC, Han Y, Kuo J. A role for antimetabolites in glaucoma tube surgery: current evidence and future directions. Curr Opin Ophthalmol. 2016 Mar;27(2):164-9. doi: 10.1097/ICU.0000000000000244. PMID 26720778
- [Background] Cui QN, Hsia YC, Lin SC, Stamper RL, Rose-Nussbaumer J, Mehta N, Porco TC, Naseri A, Han Y. Effect of mitomycin c and 5-flurouracil adjuvant therapy on the outcomes of Ahmed glaucoma valve implantation. Clin Exp Ophthalmol. 2017 Mar;45(2):128-134. doi: 10.1111/ceo.12811. Epub 2016 Sep 1. PMID 27490793
- [Background] Costa VP, Azuara-Blanco A, Netland PA, Lesk MR, Arcieri ES. Efficacy and safety of adjunctive mitomycin C during Ahmed Glaucoma Valve implantation: a prospective randomized clinical trial. Ophthalmology. 2004 Jun;111(6):1071-6. doi: 10.1016/j.ophtha.2003.09.037. PMID 15177955
- [Background] Kook MS, Yoon J, Kim J, Lee MS. Clinical results of Ahmed glaucoma valve implantation in refractory glaucoma with adjunctive mitomycin C. Ophthalmic Surg Lasers. 2000 Mar-Apr;31(2):100-6. PMID 10743919
- [Background] Tien M., Yip L., Wong E.P.Y., Yong V., Wong H.T. & Lim B.A. (2013). The effect of adjuvant mitomycin C in ahmed glaucoma valve surgery for refractory glaucoma. Investigative Ophthalmology and Visual Science, 54(15), no pagination. Retrieved from http://ovidsp.ovid.com/ovidweb.cgi?T=JS&PAGE=reference&D=emed14&NEWS=N&AN=628682336.
- [Background] Kurnaz E, Kubaloglu A, Yilmaz Y, Koytak A, Ozerturk Y. The effect of adjunctive Mitomycin C in Ahmed glaucoma valve implantation. Eur J Ophthalmol. 2005 Jan-Feb;15(1):27-31. PMID 15751236
- [Background] Bikbov MM, Khusnitdinov II. The Results of the Use of Ahmed Valve in Refractory Glaucoma Surgery. J Curr Glaucoma Pract. 2015 Sep-Dec;9(3):86-91. doi: 10.5005/jp-journals-10008-1191. Epub 2016 Feb 2. PMID 26997843
- [Background] Alvarado JA, Hollander DA, Juster RP, Lee LC. Ahmed valve implantation with adjunctive mitomycin C and 5-fluorouracil: long-term outcomes. Am J Ophthalmol. 2008 Aug;146(2):276-284. doi: 10.1016/j.ajo.2008.04.008. Epub 2008 Jun 6. PMID 18538300
- [Background] Park Y, Cho KJ. Posterior segment complications of Ahmed valve implantation. BMC Ophthalmol. 2022 Feb 15;22(1):78. doi: 10.1186/s12886-022-02297-y. PMID 35168587